CLINICAL TRIAL: NCT06247891
Title: Endocytoscopy of Upper Gastrointestinal Tract in Acute Graft-versus-host Disease: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023309
Record Dates: First submitted 2024-01-08; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Endocytoscopy
Keywords: Endocytoscopy; acute graft-versus-host disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Group (Other)
  Interventions: Procedure: ECS Group

INTERVENTIONS:
Procedure: ECS Group — Patients underwent endoscopic and endocytoscopic evaluations.

SUMMARY:
The goal of this clinical trial is to test the assess the diagnostic effectiveness of endocytoscopy in patients with underlying UGI aGvHD. The main question it aims to answer is: the effectiveness of ECS for diagnosing UGI aGvHD. Participants will undergo endoscopy, endocytoscopic evaluation and biopsy simultaneously. If there is a comparison group: Researchers will compare endoscopic, endocytoscopic and pathologic findings of these patients.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 14 years
* developed UGI symptoms within first three months after engraftment or during the tapering of immunosuppressive agents

Exclusion Criteria:

* < 14 year
* with underlying gastrointestinal disease before allo-HSCT
* incomplete medical information

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
the effectiveness of endocytoscopy for diagnosing UGI aGvHD | three months
  the percentage of esophageal, gastric, and duodenal UGI aGvHD diagnosed by endocytoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ye Zhao, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP